CLINICAL TRIAL: NCT06063889
Title: Assessment of Maximal Rate of Force Development of Ankle Muscles and Its Association Functional Ability in Patients With Knee Osteoarthritis
Brief Title: Maximal Rate of Force Development of Ankle Muscles and Functional Ability in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Director of Electromyography lab, Ahram Canadian University
Other Study IDs: 012/90002023
Record Dates: First submitted 2023-09-26; First posted 2023-10-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Knee Osteoarthritis; Knee Arthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Knee OA Patients: This group consists of patients who have been diagnosed with knee osteoarthritis. They will be subjected to a series of tests to assess the maximal rate of force development of ankle muscles and their functional abilities.
  Interventions: Diagnostic Test: Maximal Rate of Force Development Test for Ankle Muscles
- Healthy Control: This group will include healthy individuals without knee osteoarthritis. They will undergo the same series of tests to serve as a control group, enabling the comparison of results with the Knee OA Patients group.
  Interventions: Diagnostic Test: Maximal Rate of Force Development Test for Ankle Muscles

INTERVENTIONS:
Diagnostic Test: Maximal Rate of Force Development Test for Ankle Muscles — This test is designed to measure the maximal rate of force development in the ankle muscles, specifically the plantar flexors. It aims to assess the relationship between the strength of these muscles and the functional ability in patients with knee osteoarthritis. The results from this test will help to understand how lower limb muscle strength influences the symptoms and progression of knee osteoarthritis.

SUMMARY:
This study is a detailed assessment of the maximal rate of force development of ankle muscles and its association with functional ability in patients with knee osteoarthritis (OA).

DETAILED DESCRIPTION:
This research is designed to study the link between force development in ankle muscles and functional abilities in knee OA patients. It aims to understand the influence of ankle muscle strength, specifically plantar flexors, on the stability, pain, and functionality of patients with knee OA. The study will analyze the rate of force development, its importance in explosive strength improvement, and impact on preventing knee injuries. Furthermore, it will investigate the compensatory mechanism of the plantar flexors developed by patients in advanced stages to balance other muscle failures.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 (Knee OA group)

  1. Patients diagnosed with knee osteoarthritis according to Performance of the 2018 classification criteria for early stage knee OA was tested using data from the Osteoarthritis Initiative (OAI (Leung et al.,2020).
  2. Grade 2-3 KOA cases according to Kelgren-Lawrance classification
  3. Having knee pain for at least 6 months.
  4. The visual analog scale (VAS) score being at least 3 or more.
* Group 2 (Healthy control group) 1. Individuals with no signs or symptoms of Knee OA or other neurological or musculoskeletal conditions.

Exclusion Criteria:

1. Patellar subluxation
2. Surgery in any joint of the lower limb
3. Meniscal injury
4. Ligament instability
5. Patients who received intra-articular injection in the knee in the last 6 months
6. Patients with problems in the hip and ankle
7. Patients who participated in in another physical therapy program in the last 3 months were not included in the study.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients suffering from knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2023-07-20 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

PRIMARY OUTCOMES:
Knee Osteoarthritis Outcome Score (KOOS) | Baseline
  The KOOS is a questionnaire that assesses five aspects of knee injury and osteoarthritis: pain, symptoms, ADL function, sport and recreation function, and quality of life. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems. Higher scores indicate better function and less pain.
Forward Step Down Test (FSDT) | Baseline
  This functional ability test requires participants to perform as many repetitions as possible in 30 seconds of a specific movement. The number of valid repetitions performed in this duration is recorded.
Single Leg Hop Test (SLHT) | Baseline
  n this test, participants hop forward as far as possible on one leg, and the distance hopped is recorded.
Isokinetic Testing Procedures | Baseline
  This procedure involves conducting tests of three (60°/s) or five (120°/s) maximal nonconsecutive efforts with specific rest intervals. Each subject is instructed to exert maximal effort throughout the whole range of motion.
Rate of Force Development (RFD) | Baseline
  The RFD is a measure of the speed at which the force of a muscle contraction develops. It is typically measured during isometric contractions and provides information about the muscle's explosive strength capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Abdelrahman, Ph.D, Study Chair — Cairo University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No